CLINICAL TRIAL: NCT06377202
Title: Long-Term Follow-Up Safety Study of Subjects Treated with SynKIR-110, Autologous T Cells Transduced with Mesothelin KIR-CAR, in Cancer Studies
Brief Title: Long-Term Follow-Up Safety Study of Subjects Treated with SynKIR-110 in Cancer Studies
Status: Withdrawn | Type: Observational
Why Stopped: The study is being withdrawn and replaced by a new multicenter LTFU Basket Study, designed to monitor the long-term safety of all SynKIR CAR T cell products. This updated study will include all participants who have been treated with Verismo Therapeu
Sponsor: Verismo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: SynKIR-110 LTFU
Record Dates: First submitted 2024-04-10; First posted 2024-04-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC (RCL-VSV-G) Whole Blood (qPCR persistence)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of SynKIR- 110 administered to adult subjects with solid tumors expressing mesothelin.

DETAILED DESCRIPTION:
This study has been designed in adherence with the following Food and Drug Administration (FDA) Guidance documents for Industry: the January 2020 Long-Term Follow-Up After Administration of Human Gene Therapy Products; the January 2020 Testing of Retroviral Vector-Based Human Gene Therapy Products for Replication Competent Retrovirus During Product Manufacture and Patient Follow-up; and the March 2022 Considerations for the Development of Chimeric Antigen Receptor (CAR) T Cell Products. The study serves to collect data on delayed adverse events for up to fifteen (15) years following a single infusion of SynKIR-110 administered to advance cancer patients with mesothelin expressing tumors.

For subjects who have not progressed and have rolled onto this LTFU study at 12 months, data on long-term clinical activity will be collected from the subject's standard of care treatment/medical records.

Safety monitoring for delayed adverse events related to SynKIR-110 will include physical examinations, laboratory assessments including complete blood counts, complete metabolic profile, RCL testing and testing for persistence of lentiviral mediated T cells.

Testing for persistence of vector sequences by PCR in subjects' blood (and possibly other surrogate tissue) samples will be done at intervals no greater than 6 months for the first five years and then no greater than annually for the next 10 years, or until such time that no vector sequences are detectable in the subjects' sample.

Subject samples will be collected for RCL (qPCR for VSV-G) assessment at 3, 6, and 12 months after SynKIR-110 infusion and yearly for up to fifteen (15) years. If all RCL tests within the first year are negative for an individual patient, collection of the yearly follow-up samples may be discontinued for that individual.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have received any amount of SynKIR-110 in a study sponsored by Verismo Therapeutics.
2. Adult 18 years of age or older

Exclusion Criteria:

1. Unable or unwilling to provide written informed consent
2. Unable or unwilling to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who recieved SynKIR-110
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2038-12-15 (Estimated); Study Completion 2038-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment related adverse events as assessed by CTCAE v5.0 | 15 years from date subject received SynKIR-110
  Monitor for signs of SynKIR-110 related delayed adverse events

SECONDARY OUTCOMES:
Number of subjects with persistence of SynKIR-110 modified cells | 15 years from date subject received SynKIR-110
  Monitor qPCR of peripheral blood for persistence of SynKIR-110 modified T cells.
Number of subjects with potential/suspected RCL | 15 years from date subject received SynKIR-110
  Monitor qPCR of peripheral blood for VSV-G DNA

CONTACTS AND LOCATIONS:
Overall Officials: Laura Johnson, PhD, Study Director — Verismo Therapeutics
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No